CLINICAL TRIAL: NCT01604447
Title: Randomized Evaluation of the Use of Plastic Bags to Prevent Neonatal Hypothermia in Developing Countries-Part IV
Brief Title: Evaluation of Use of Plastic Bags to Prevent Neonatal Hypothermia-Part IV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Children's of Alabama (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UAB Neo 009
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-02

CONDITIONS: Hypothermia
Keywords: Hypothermia; Newborn; Incubator; Plastic bag; Normothermia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Incubator removal-torso bag (Active Comparator): Use plastic bag covering the torso and lower extremities for temperature regulation with standard bundling practices when removing infant from incubator
  Interventions: Procedure: Hypothermia prevention with plastic bag
- Incubator removal-no plastic bag (Placebo Comparator): Standard bundling practices when removing the infant from the incubator. No plastic bag used.
  Interventions: Procedure: Hypothermia prevention without plastic bag

INTERVENTIONS:
Procedure: Hypothermia prevention with plastic bag — Upon removal from the incubator, infant will be placed into a plastic bag to his/her axillae, and the bag will be folded and taped to itself to prevent it from covering the infant's nose or mouth. The infant will be wrapped in a blanket and receive a cloth hat. The bag will be changed when soiled and the infant will remain in the bag for 72 hours or until discharge, whichever comes first. The infant's temperature will be monitored for 72 hours or until discharge, whichever comes first.
  Arms: Incubator removal-torso bag
Procedure: Hypothermia prevention without plastic bag — Upon removal from incubator, the infant will be wrapped in a blanket and receive a cloth hat, according to standard bundling practices. The infant's temperature will be monitored for 72 hours or until discharge, whichever comes first.
  Arms: Incubator removal-no plastic bag

SUMMARY:
The overall hypothesis is that plastic bags used in combination with WHO thermoregulation care will reduce the incidence of hypothermia in preterm/low birth weight and full term infants when compared to routine WHO thermoregulation care alone. Part V is comparing use of a plastic torso wrap to no plastic torso wrap in preterm/low birth weight infants following removal from their incubator to assist with temperature regulation.

DETAILED DESCRIPTION:
Due to limited resources and numbers of incubators, hospitals in developing countries remove infants from incubators at lower weights than in developed countries, putting infants at increased risk for hypothermia. This study will compare the incidence of hypothermia during the 72 hours after incubator removal of infants randomized to receive standard incubator removal (control group) or standard incubator removal with a plastic bag covering their torsos and lower extremities (intervention group). The axillary temperature of each infant will be taken upon removal from the incubator, every subsequent 6-8 hours, and finally, at 72 hours as the bags are removed. Blood pressure, blood sugar, seizures, weight gain, hyperthermia, death, observation for respiratory distress, bronchopulmonary dysplasia, sepsis, intraventricular hemorrhage, periventricular leukomalacia, necrotizing enterocolitis, intestinal perforation, pulmonary hemorrhage room temperature and humidity, and length of time in an incubator will be recorded throughout their hospitalization for all infants. With an estimated hypothermia incidence of 30% and a hypothesized 20% absolute risk reduction (66% relative risk reduction), a sample size of 118 will be used to have a power of 80% and a confidence interval of 95%.

ELIGIBILITY:
Inclusion Criteria:

* Infant admitted to the NICU
* Current weight less than 2,000g
* Being removed from incubator

Exclusion Criteria:

* Abdominal wall defect or myelomeningocele
* Major congenital anomalies
* Blistering skin disorder

Ages: 1 Hour to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 118 (Actual)
Dates: Start 2012-06; Primary Completion 2014-08 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Axillary temperature 36.5-37.5 degrees Celsius | 1-72 hours
  Temperature taken per axilla for one minute

SECONDARY OUTCOMES:
Blood pressure | Up to 4 weeks
  Measure of extremity blood pressure per cuff taken during nursery stay
Blood glucose | Up to 4 weeks
  Measure of blood glucose per laboratory value taken per heel stick
Seizure | Up to 4 weeks
  Seizure activity diagnosed by medical doctor or nurse. No electoencephalogram will be done.
Weight gain | Up to 4 weeks
  Infant will be weighed daily and rates of weight gain will be calculated
Respiratory Distress Syndrome (RDS) | Up to 4 weeks
  Documentation of increased work of breathing, retractions, and a need for oxygen, intubation, or surfactant
Bronchopulmonary Dysplasia (BPD) | 28 days after birth
  Oxygen requirement at 28 days of life
Pneumothorax | Up to 4 weeks
  Either chest radiograph documentation or clinical deterioration consistent with air leak
Sepsis | Up to 4 weeks
  Culture proven or culture negative clinically treated course consistent with sepsis
Major brain injury | Up to 4 weeks
  Intracranial hemorrhage grade 3-4 or periventricular leukomalacia documented on cranial ultrasound
Necrotizing enterocolitis or intestinal perforation | Up to 4 weeks
  Documentation of pneumatosis or intestinal perforation on x-ray or treatment course for clinical necrotizing enterocolitis per Bell's Classification stage greater than 1.
Pulmonary hemorrhage | Up to 4 weeks
  Blood seen in the endotracheal tube and treated by physician
Death | Up to 4 weeks
  Cardiorespiratory failure
Hyperthermia | Up to 4 weeks
  Axillary temperature > 38 degrees Celsius per temperature taken per axilla for 1 minute
Length of time in incubator | Up to 4 weeks
  Documentation of length of time spent in incubator and number of times placed in incubator
Room temperature and humidity | 1-72 hours
  A recording of the room temperature and humidity will be obtained with each axillary temperature measurement
Incubator temperature and humidity | 1 hour
  A recording of the air temperature and humidity with the incubator will be obtained with each axillary temperature measurement

CONTACTS AND LOCATIONS:
Overall Officials: Waldemar A Carlo, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University Teaching Hospital, Lusaka, Zambia